CLINICAL TRIAL: NCT02700113
Title: Investigating Phenotypic Profiles of Minimally Verbal Children and Adolescents With ASD/Profiles of Abilities in Children and Adolescents With ASD
Brief Title: Investigating Phenotypic Profiles of Children and Adolescents With ASD
Acronym: Phenotyping
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Northeastern University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Helen B. Tager-Flusberg, Professor, Boston University
Other Study IDs: 3646E; P50DC013027 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ASD: There is only one group; minimally verbal individuals with Autism Spectrum Disorder aged 4 to 17 years.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Intervention is not a part of this study. This is a behavioral phenotyping study of minimally verbal individuals with Autism Spectrum Disorder.

SUMMARY:
The purpose of this study is to provide a detailed description of language and cognitive profiles found among children and adolescents diagnosed with autism spectrum disorders (ASD). Participants with ASD ages 4-17;12 years who have limited verbal skills will be given comprehensive behavioral assessments to collect data that will advance our understanding of language-related processes in individuals with ASD, the knowledge of which will help in designing future interventions for this population.

DETAILED DESCRIPTION:
About 25% to 30% of children with ASD fail to acquire spoken language. This group of children and adolescents with ASD has been neglected in research conducted over the past 2 decades, in part because the field lacks the tools to assess them, and they often pose significant behavioral challenges that preclude their participation in research studies. Among the ~70% individuals with ASD who have spoken language skills, about 50% are language impaired; the remaining group have normal language scores on standardized tests. To date, studies of brain and cognitive mechanisms that underlie this heterogeneity in ASD remain limited. The goal of this study, which is part of the Autism Center of Excellence, is to provide a detailed description of phenotypic profiles found among minimally verbal individuals diagnosed with ASD. Participants with ASD ages 4 to 18 will be given comprehensive assessments, including standardized assessments of language, nonverbal cognitive abilities and adaptive functioning. Assessments will also include experimental tasks based on using eye-tracking, touch screen and electrophysiology technology (EEG), parent-report measures and parent-child interaction measures. The eye-tracking and touch screen assessments will target receptive language, word learning mechanisms, and social attention deployment to visual and auditory stimuli. The EEG/ERP assessments will target auditory processing and organization, with specific focus on mismatch negativity (MMN) markers of auditory processing. Based on these comprehensive assessments the investigators aim to generate a description of the cognitive-behavioral phenotypes common to minimally verbal autistic individuals. The investigators will also investigate age-related patterns in the development of behavioral phenotypes and the role of symptom severity in shaping phenotypic profiles in this population. The investigators expect that their findings will provide valuable insights into the etiology of profound expressive language deficits in a significant proportion of the ASD population and will lead to identifying subphenotypes within the minimally verbal population.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they have a formal diagnosis of ASD, are 4-18 years old, and have a very small repertoire of spoken words or fixed phrases that are used communicatively, and that are restricted to limited contexts and functions (e.g. requests with familiar adults).

Exclusion Criteria:

* have a history of significant neurological diseases, TBI, sensory impairment (e.g., significant visual or hearing impairment)
* English is not the primary language spoken in the household.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2019-06 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Autism Spectrum Diagnosis | 5 years
  Interview
Adaptive Abilities | 5 years
  Interview
Cognitive Abilities | 5 years
  Interview
Language | 5 years
  Interview
Social Behavior | 5 years
  Interview
Repetitive Behavior | 5 years
  Questionnaire
Sensory Behaviors | 5 years
  Questionnaire
Atypical Behavior | 5 years
  Questionnaire
Psychopathology | 5 years
  Questionnaire
Emotion Regulation | 5 years
  Questionnaire
Handedness | 5 years
  Questionnaire
Electrophysiological Measures and Neural Oscillatory Patterns of Perception, Organization, and Analysis of Auditory scenes | 5 years
  Physiological parameter
Indices of social attention deployment measured by unobtrusively recording participants' eye-movements during the passive viewing of brief realistic video-clips. | 5 years
  Physiological parameter
Indices of electrodermal activity (EDA) measured wirelessly with the Q sensor (a small wearable device designed to work in real-world environments in an untethered, unobtrusive way). | 5 years
  Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Helen Tager-Flusberg, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tager-Flusberg H, Kasari C. Minimally verbal school-aged children with autism spectrum disorder: the neglected end of the spectrum. Autism Res. 2013 Dec;6(6):468-78. doi: 10.1002/aur.1329. Epub 2013 Oct 7. PMID 24124067
- See also: This is the website for our center. — http://www.bu.edu/autism